CLINICAL TRIAL: NCT03080363
Title: Is Painless ESWL Possible? Analgesic Efficacy of Ultrasound Guided Quadratus Lumborum Block During Extracorporeal Shockwave Lithotripsy
Brief Title: Analgesic Efficacy of Ultrasound Guided Quadratus Lumborum Block During ESWL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ataturk University ESWL
Record Dates: First submitted 2017-03-06; First posted 2017-03-15 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Pain, Acute
Keywords: Extracorporeal Shockwave Lithotripsy; Quadratus Lumborum Block; bupivacaine; lidocaine
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (Active Comparator): Ultrasound guided Quadratus Lumborum Block with 10 ml %0.5 bupivacaine and 10 ml %2 lidocaine
  Interventions: Drug: Bupivacaine; Drug: Lidocaine
- Group Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Bupivacaine — 10 ml %0.5 bupivacaine
  Arms: Quadratus Lumborum Block
Drug: Lidocaine — 10 ml %2 lidocaine
  Arms: Quadratus Lumborum Block

SUMMARY:
Extracorporeal shockwave lithotripsy (ESWL) is widely used for the treatment of urinary tract calculi; however, the vast majority of patients do not tolerate the procedure without analgesia and sedation.

Lots of methods have been tried to control this pain (non-steroidal anti-inflammatory drugs, opioids, alpha 2 agonists, transversus abdominis plane block with long-acting local anesthetics, paravertebral block, local anesthetics infiltration, lidocaine/prilocaine cream).

The quadratus lumborum block was first described by Blanco. QL block is performed as one of the perioperative pain management procedures for abdominal surgery. QL block provides anesthesia and analgesia on the anterior and lateral wall of the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II patients undergoing Extracorporeal Shockwave Lithotripsy

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Score | Intraoperative 30 minutes
  Visual Analog Pain Score at 5.,10.,15., 20., 25., 30. minutes

SECONDARY OUTCOMES:
Opioid consumption | Intraoperative 30 minutes
  Opioid consumption at 5.,10.,15., 20., 25., 30. minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elnabtity AM, Tawfeek MM, Keera AA, Badran YA. Is unilateral transversus abdominis plane block an analgesic alternative for ureteric shock wave lithotripsy? Anesth Essays Res. 2015 Jan-Apr;9(1):51-6. doi: 10.4103/0259-1162.150177. PMID 25886421
- [Background] Hanoura S, Elsayed M, Eldegwy M, Elsayed A, Ewieda T, Shehab M. Paravertebral block is a proper alternative anesthesia for outpatient lithotripsy. Anesth Essays Res. 2013 Sep-Dec;7(3):365-70. doi: 10.4103/0259-1162.123238. PMID 25885985